CLINICAL TRIAL: NCT02408159
Title: A Double Blind Placebo-controlled Randomized Study of Varicella Zoster Vaccine in Patients With Moderate-to-severe Plaque Psoriasis Who Are Candidates for Biologic Therapy
Brief Title: Varicella Zoster Vaccine in Patients With Plaque Psoriasis Treated With Biologic Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Inno-6041
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-08

CONDITIONS: Psoriasis
Keywords: Live, attenuated virus varicella-zoster vaccine; Zostavax; herpes zoster; shingles
MeSH Terms: conditions — Psoriasis; Herpes Zoster | interventions — Herpes Zoster Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varicella Zoster Vaccine (Experimental): Sterile, lyophilized white to off-white compact crystalline plug in a single-dose vial. Each vial contains one dose of lyophilized vaccine (approximately 0.65 mL when reconstituted as directed). The diluent (0.7 mL) is a sterile, clear, colorless fluid supplied separately in a 3 mL single-dose vial. A single dose will be administered to subjects at baseline.
  Interventions: Drug: Varicella Zoster Vaccine
- 0.9% Sodium Chloride (Placebo Comparator): United States Pharmacopeia (USP), preservative free for injection supplied in a single dose vial.
  A single dose will be administered to subjects at baseline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varicella Zoster Vaccine
  Other Names: Zostavax®
  Arms: Varicella Zoster Vaccine
Drug: Placebo
  Other Names: 0.9% Sodium Chloride; Saline 0.9%
  Arms: 0.9% Sodium Chloride

SUMMARY:
This study will evaluate the ability of the vaccine to produce antibodies against herpes zoster virus (shingles) and safety of vaccination with Varicella Zoster Vaccine in patients with moderate to severe psoriasis who will initiate biologic therapy 4 to 6 weeks after vaccination.

Varicella Zoster Vaccine will be administered 4 to 6 weeks prior to receipt of biological therapy and will be compared against placebo.

This double-blind study will enroll approximately 50 adult patients with moderate-to-severe plaque psoriasis in approximately 3 centers in Canada. Study products will be assigned randomly at a 4:1 ratio.

For each patient who is included, the study may last up to 22 weeks, including the screening and the follow-up period. During the study, subjects will come to the dermatology clinic up to 4 occasions: for a screening visit, Baseline visit, Day 42 as well as 84 days after they started taking the biological treatment for a last visit. If patients develop a varicella-like or shingles-like rash at any time after they received the vaccine, they will be requested to come back to the clinic within 72 hours of rash onset (preferably within 24 hours) for examination. Subjects will be asked to provide a lesion swab/vesicular fluid in this case.

ELIGIBILITY:
Main Inclusion Criteria:

1. Outpatient men or women aged 50 years or older
2. Must have moderate-to-severe plaque psoriasis for at least 6 months, and for whom a decision to use biologic therapy has been made, with biologic therapy planned to be initiated within the next 4-6 weeks.
3. History of varicella, or having resided in Canada for at least 30 years.

Main Exclusion Criteria:

1. Have received Varicella Zoster Vaccine vaccine or known allergies to the Varicella Zoster Vaccine vaccine or its excipients including neomycin and gelatin
2. Primary and acquired immunodeficiency states due to conditions such as: acute and chronic leukemias, lymphoma, other conditions affecting the bone marrow or lymphatic system, immunosuppression due to HIV/AIDS, cellular immune deficiencies.
3. Current use of non-topical antiviral therapy with known activity against varicella-zoster virus.
4. Exposure to varicella or zoster within 28 days prior to vaccination.
5. Patients who are diagnosed with herpes zoster at the time of the vaccination.
6. Active untreated tuberculosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Varicella Zoster Virus (VZV) antibody | 42 Days
  Geometric mean several fold rise in Varicella Zoster Virus (VZV) antibody from baseline to Day 42 as measured by glycoprotein-based enzyme-linked immunosorbent assay (gpELISA)

SECONDARY OUTCOMES:
Geometric mean titer of VZV antibody | 42 Days
  Change from baseline in geometric mean titer of VZV antibody at Day 42 as measured with gpELISA.
Serious Adverse Events | 84 Days
  Proportion of patients randomized to Varicella Zoster Vaccine presenting vaccine related serious adverse events (SAEs) during the study as compared to patients randomized to placebo.
Presenting with Varicella or Herpes Zoster | 84 Days
  Proportion of patients randomized to Varicella Zoster Vaccine presenting varicella or herpes zoster during the study as compared to patients randomized to placebo

OTHER OUTCOMES:
Psoriasis Area Severity Index (PASI) | 84 Days
  Change from baseline in Psoriasis Area Severity Index (PASI) at Day 84 post-biologic in patients randomized to Varicella Zoster Vaccine as compared to patients randomized to placebo.
Body Surface Area (BSA) | 84 Days
  Change from baseline in Body Surface Area (BSA) at Day 84 post-biologic in patients randomized to Varicella Zoster Vaccine as compared to patients randomized to placebo.
Physician Global Assessment (PGA) | 84 Days
  Change from baseline in Physician Global Assessment (PGA) at Day 84 post-biologic in patients randomized to Varicella Zoster Vaccine as compared to patients randomized to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Guenther, MD, FRCPC, Principal Investigator — The Guenther Dermatology Research Center
Locations (3):
- Canada (3):
  - Inno-6041 study site, London, Ontario
  - Inno-6041 study site, Markham, Ontario
  - Innovaderm Research Inc., Montreal, Quebec